CLINICAL TRIAL: NCT03019120
Title: The Effect of Vitamin D Supplementation on Neurocognitive Function in Older Subjects
Brief Title: Vitamin D Supplementation and Neurocognition
Acronym: Dcog
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to administrative reasons, it was not possible to enroll subjects.
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Tzvi Dwolatzky, Prof., Rambam Health Care Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0103-16-LND
Record Dates: First submitted 2017-01-09; First posted 2017-01-12 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Vitamin D Deficiency; Neurocognitive Dysfunction
MeSH Terms: conditions — Vitamin D Deficiency; Cognition Disorders | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Comparator: Intervention group (Experimental): Vitamin D supplementation for subjects with below normal levels of this vitamin.
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — 1. Subjects will undergo a cognitive evaluation using the Montreal Cognitive Assessment (MoCA) screening test and the Neurotrax computerized cognitive assessment battery.
  2. Subjects will receive a supplemental monthly oral dose of 60000 units Vitamin D administered by a nurse for a period of 3 months.
  3. Levels of serum calcium will be repeated monthly (end of month 1, 2, 3).
  4. Subjects will undergo a repeat blood test to examine the level of vitamin D at the end of 3 months of follow-up.
  5. At 3-month follow-up subjects will be asked to complete the Neurotrax computerized cognitive assessment battery.

SUMMARY:
This study will evaluate the effect of vitamin D supplementation on the neurocognitive function of older people with lower than normal levels of vitamin D at baseline

DETAILED DESCRIPTION:
Background: Ageing is associated with an increased risk of cognitive decline. Vitamin D plays an important role in many of the symptoms and conditions related to advanced age, including impaired balance, falls and osteoporosis. Vitamin D also has a physiological effect on the function of the central nervous system, and studies have suggested a relationship between this vitamin and changes in cognitive function of older people. The investigators propose a pilot study to evaluate the effect of vitamin D supplementation on the neurocognitive function of older people.

Methods: A total of 30 subjects of both genders older than 65 years with levels of 25-OH Vitamin D lower than 30 ng/ml on routine laboratory screening will be included in the study. Exclusion criteria will include any unstable medical condition as determined by the treating physician, a diagnosis of dementia, the use of supplements containing vitamin D in any dose, significant visual or hearing impairment not corrected by spectacles or hearing aids, and a level of literacy that limits the performance of computerized neurocognitive testing. Following provision of written informed consent for inclusion in the study, subjects will answer a questionnaire providing demographic details, undergo cognitive screening by use of the MoCA test, and computerized cognitive assessment using the Neurotrax battery. All subjects will undergo repeat testing for level of 25-OH Vitamin D, and where below-normal levels are confirmed patients will receive a supplemental monthly oral dose of 60000 units Vitamin D administered by a nurse for a period of 3 months. Levels of serum calcium will be repeated monthly (end of month 1, 2, 3). At 3 months subjects will undergo repeat testing for level of 25-OH Vitamin D, and repeat computerized cognitive assessment using the Neurotrax battery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 years and older.
* Level of vitamin D (25-OH vitamin D) is less than 30 ng / ml.
* Stable health status as assessed by the treating primary care physician.
* Do not take supplements containing vitamin D.
* Normal cognitive function as determined by MoCA Test screening and clinical assessment
* Adequate literacy to enable the performance of cognitive assessment instruments
* Provide informed consent as required by the Ethics Committee.

Exclusion Criteria:

* Age younger than 65 years
* Health status not stable as determined by the treating primary care physician
* A diagnosis of dementia
* Taking supplements containing Vitamin D
* Significant visual or hearing impairment not corrected by spectacles or hearing aids
* Impaired competency limiting the subject's ability to provide informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function as assessed by the Neurotrax computerized cognitive assessment battery | 3 months
  The Neurotrax computerized cognitive assessment instrument measures the following domains: Memory, executive functions, attention, verbal functions and motor skills. This instrument was found to have high validity in identifying patients who suffer from cognitive decline in comparison to healthy patients in the elderly. There are many advantages to a computerized cognitive assessment tool. It allows a measurement of various cognitive domains as well as an accurate, detailed and objective measurements of patients. It is also very sensitive to cognitive changes occurring in a specific individual over time.

CONTACTS AND LOCATIONS:
Overall Officials: Elad Rubin, M.A, Study Director — Rambam Health Care Campus
Locations (1):
- Laniado Medical Center, Netanya, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Annweiler C, Allali G, Allain P, Bridenbaugh S, Schott AM, Kressig RW, Beauchet O. Vitamin D and cognitive performance in adults: a systematic review. Eur J Neurol. 2009 Oct;16(10):1083-9. doi: 10.1111/j.1468-1331.2009.02755.x. Epub 2009 Jul 29. PMID 19659751
- [Background] Buell JS, Dawson-Hughes B. Vitamin D and neurocognitive dysfunction: preventing "D"ecline? Mol Aspects Med. 2008 Dec;29(6):415-22. doi: 10.1016/j.mam.2008.05.001. Epub 2008 May 13. PMID 18579197
- [Background] Dwolatzky T, Whitehead V, Doniger GM, Simon ES, Schweiger A, Jaffe D, Chertkow H. Validity of a novel computerized cognitive battery for mild cognitive impairment. BMC Geriatr. 2003 Nov 2;3:4. doi: 10.1186/1471-2318-3-4. PMID 14594456
- [Background] Lifshitz M, Dwolatzky T, Press Y. Validation of the Hebrew version of the MoCA test as a screening instrument for the early detection of mild cognitive impairment in elderly individuals. J Geriatr Psychiatry Neurol. 2012 Sep;25(3):155-61. doi: 10.1177/0891988712457047. PMID 23124009